CLINICAL TRIAL: NCT01714180
Title: Effect of Body Mass on Acyclovir Pharmacokinetics
Status: Completed | Type: Observational
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Aaron Cumpston, PharmD, Pharmacy Clinical Specialist - BMT/Hematologic Malignancy, West Virginia University
Other Study IDs: WVU 031112; 24368 (Other: West Virginia University IRB)
Record Dates: First submitted 2012-10-17; First posted 2012-10-25 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Hematological Malignancy; Pharmacokinetics of Acyclovir
Keywords: Acyclovir; Pharmacokinetics; Obese; Non-obese; Weight; Distribution; Clearance
MeSH Terms: conditions — Hematologic Neoplasms; Obesity; Body Weight

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Obese Patients
- Non-obese Patients

SUMMARY:
Studies have shown that different percentages of body fat can alter the way drugs are distributed in the body. This study will use blood samples taken at different time points for patients taking acyclovir to determine if higher body weights affect drug exposure. The information gathered from this study will help understand if patients with higher body weights need a different dosing plan.

Patients receiving acyclovir as standard of care will be enrolled into this study. They will have blood draws once before they take acyclovir and 10 times after they take the acyclovir (over a total of 12 hours). These patients will be in the hospital already and will not need to make additional trips back to have blood drawn. A total of about 4-5 tablespoons of blood will be drawn for this study. 7 obese patients and 7 matched, non-obese patients will be enrolled into this study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years of age
* Receiving intravenous acyclovir 5 mg/kg (total body weight [TBW] for normal weight patients and ideal body weight [IBW] for obese patients) as part of their routine care
* Admitted as an inpatient with an expected stay of at least 24 hours
* Weight > 190% of ideal body weight (IBW) for "obese" patients or weight 80-120% of IBW for matched control patients.

Exclusion Criteria:

* Receipt of acyclovir or similar agents (valacyclovir, ganciclovir, valganciclovir, famciclovir) in the prior 24 hours
* Serum creatinine > 1.5 mg/dL at time of drug administration
* Hypersensitivity to acyclovir
* Patients requiring ventilator support or vasopressors in the prior 24 hours
* Receipt of probenecid, mycophenolate, tenofovir, or zidovudine in the prior 7 days
* Pregnant or breast-feeding
* Significant anatomical deformities that influence body habitus (i.e. amputation)
* Prior inclusion in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese and normal weight patients treated with acyclovir in an inpatient setting.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2012-10; Primary Completion 2014-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Systemic clearance of acyclovir in obese and non-obese patients | 12 hours after acyclovir dose

SECONDARY OUTCOMES:
Alpha and beta half-life of acyclovir in obese and non-obese patients | 12 hours after acyclovir dose
Maximum concentration (Cmax) of acyclovir in obese and non-obese patients | 12 hours after acyclovir dose
Time to maximum concentration (Tmax) of acyclovir in obese and non-obese patients | 12 hours after acyclovir dose
Volume of distribution (Vd and Vdss) of acyclovir in obese and non-obese patients | 12 hours after acyclovir dose
Time that concentration is above IC50 for varicella and herpes viruses 4,5,6,7 for acyclovir in obese and non-obese patients | 12 hours after acyclovir dose

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Cumpston, PharmD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University Hospitals Mary Babb Randolph Cancer Center, Morgantown, West Virginia, United States

REFERENCES:
- [Derived] Turner RB, Cumpston A, Sweet M, Briggs F, Slain D, Wen S, Craig M, Hamadani M, Petros W. Prospective, Controlled Study of Acyclovir Pharmacokinetics in Obese Patients. Antimicrob Agents Chemother. 2016 Jan 11;60(3):1830-3. doi: 10.1128/AAC.02010-15. PMID 26824940